CLINICAL TRIAL: NCT00125411
Title: Phase I Study of the Oral Platinum Agent Satraplatin (JM-216) in Combination With Docetaxel in Treatment of Advanced Malignancies
Brief Title: Study of Satraplatin (JM-216) in Combination With Docetaxel
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decided to discontinue study drug development.
Sponsor: Agennix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO 04904
Record Dates: First submitted 2005-07-28; First posted 2005-08-01 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Tumors
Keywords: satraplatin; docetaxel; cancer; Phase I; advanced solid tumors
MeSH Terms: conditions — Neoplasms | interventions — satraplatin; Docetaxel

INTERVENTIONS:
Drug: satraplatin and docetaxel — Satraplatin - oral administration within 2 hours of docetaxel infusion. Subsequent dosing will be on days 2-5 at approximate 24 hour intervals.
  Docetaxel will be administered as intravenous infusion over 1 hour followed by saline flush.

SUMMARY:
This is a single center, open-label, non-randomized, Phase I dose finding study of the investigational, oral cytotoxic drug, satraplatin (JM-216), in combination with docetaxel in patients with advanced solid tumors for whom curative therapy is not available. Please refer to the Eligibility Criteria below for key inclusion and exclusion criteria.

PURPOSE: The purpose of this trial is to determine a tolerable dose and schedule for the combination of satraplatin and docetaxel when given to patients with advanced solid tumors.

WHAT IS SATRAPLATIN: Satraplatin is an oral, investigational anticancer drug that is a member of the platinum-based class of chemotherapy drugs. Platinum-based drugs have been clinically proven to be one of the most effective classes of anticancer therapies. Unlike the currently marketed platinum-based drugs, satraplatin can be given orally.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignancy that is metastatic or unresectable and for which standard curative or palliative chemotherapy measures do not exist or are no longer effective
* Life expectancy of at least 3 months
* Measurable or evaluable disease
* ECOG performance status of <= 2
* Willingness and ability to give informed consent

Exclusion Criteria:

* Women who are pregnant or breastfeeding
* Other chemotherapy treatment less than 4 weeks prior to enrollment
* Treatment with docetaxel or a platinum agent less than 3 months prior to enrollment
* Other concurrent chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered investigational

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-03; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose and Safety | 3 weeks

SECONDARY OUTCOMES:
Objective response rate | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: George Wilding, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin, United States